CLINICAL TRIAL: NCT01200251
Title: The Role of Bimatoprost Eyelash Gel in Chemotherapy-induced Madarosis: an Analysis of Efficacy and Safety
Brief Title: Study of Bimatoprost Gel on Eyelash Growth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 9459; 71320 (Registry Identifier: IND)
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2010-09

CONDITIONS: Madarosis; Hypotrichosis
MeSH Terms: conditions — Hypotrichosis | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bimatoprost treated eyelid (Experimental): one eyelid of the patient was randomized to the treatment arm and given the gel to use
  Interventions: Drug: Bimatoprost eyelash gel
- control arm - no gel (No Intervention): the other fellow eyelid of the patient did not receive any treatment until month 4 and the patient crossed over to treating both eyelids

INTERVENTIONS:
Drug: Bimatoprost eyelash gel — Bimatoprost 0.03% solution was compounded into a gel - patients used on eyelash margin once daily placing gel with a fingertip or Q-tip for 6 months
  Other Names: lumigan
  Arms: Bimatoprost treated eyelid

SUMMARY:
A internally controlled, single-blinded, randomized controlled trial to investigate the use of Bimatoprost eyelash gel on eyelash growth and appearance in breast cancer patients who suffer from madarosis (loss of eyelashes) due to the side effects of chemotherapy. IND and IRB approval have been obtained.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 YO females
* madarosis or hypotrichosis (loss of eyelashes) due to chemotherapy used to treat breast cancer
* only breast cancer patients

Exclusion Criteria:

* inability to follow up, apply gel
* active eye/eyelid infection or inflammatory process
* cancer not related to breast cancer, healthy patients
* males

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2007-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
eyelash length | 6 months
  eyelash ruler used to measure eyelash length

SECONDARY OUTCOMES:
eyelash pigment | 6 mos
  blinded grader used digital photos to grade degree of pigment on scale of 1-5
eyelash thickness | 6 mos
  blinded grader used digital photos to grade degree of thickness on scale of 1-5
eyelash amount | 6 mos
  blinded grader used digital photos to grade degree of amount by counting lashes
eyelash side effects | 6 mos
  any side effects (irritation, allergy, iop change, visual acuity, macular edema, uveitis, iris color change, etc... were assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Tosti A, Pazzaglia M, Voudouris S, Tosti G. Hypertrichosis of the eyelashes caused by bimatoprost. J Am Acad Dermatol. 2004 Nov;51(5 Suppl):S149-50. doi: 10.1016/j.jaad.2004.05.002. PMID 15577756